CLINICAL TRIAL: NCT05873842
Title: TRAns-Femoral Access Intravascular Lithotripsy Comparison With PTA in TAVI
Acronym: TRAFIC-PTA
Status: Recruiting | Type: Observational
Sponsor: Rede Optimus Hospitalar SA (Network)
Responsible Party: Sponsor
Other Study IDs: RO-230301
Record Dates: First submitted 2023-05-15; First posted 2023-05-24 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Trans-femoral TAVI With Calcified Ilio-femoral Arteries
Keywords: TAVI; Calcification; Ilio-femoral arteries
MeSH Terms: conditions — Calcinosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PTA-assisted group
  Interventions: Device: Trans-femoral TAVI
- IVL-assisted group
  Interventions: Device: Trans-femoral TAVI

INTERVENTIONS:
Device: Trans-femoral TAVI — Trans-femoral TAVI (Trans-catheter Aortic Valve Implantation) with calcified ilio-femoral arteries via PTA (Percutaneous transluminal angioplasty ) or IVL (Intra-vascular Lithotripsy)

SUMMARY:
To compare the effectiveness and the safety of femoral-iliac IVL versus balloon only PTA for successful deployment of transfemoral transcatheter aortic valve prosthesis.

DETAILED DESCRIPTION:
Trans-femoral (TF) access has been identified as the best vascular approach for trans-catheter aortic valve implantation (TAVI) in the most recent European Guidelines for the treatment of valvular heart disease. Nevertheless, the TF approach is not possible in a substantial number of TAVI candidates, mainly due to the presence of important peripheral arterial disease (PAD) that is perceived as a contraindication. The presence of PAD limiting TF-TAVI feasibility has always remained a challenging scenario. The concept of preparing TF access through balloon dilatation in case of PAD had been developed and, in this context, percutaneous transluminal angioplasty (PTA) with plain-balloon has been investigated, although available literature is scarce. Intra-vascular lithotripsy (IVL) was proved effective and safe to treat calcified peripheral arteries and such new technology bares the potential for being applied in TF TAVI in patients with concomitant PAD. The rationale is that the Shockwave IVL balloon inflated at low pressure modifies the vessel rigidity with creation of multiple longitudinal and transversal cracks in the calcium present within the vessel wall. Thus, the improved vessel compliance facilitates the successful passage of the valve delivery system resulting in higher rates of procedural success and lower risk for crossover to surgery, vessel injury and major complications.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Written informed consent
3. Diagnosis of symptomatic severe aortic stenosis
4. Patient undergoing TAVI according to local institutional protocol and following Heart Team discussion.
5. High-quality Contrast-enhanced ECG gated computed tomography (CT) scan of the heart, aorta and low-limb arteries
6. Calcific severe PAD raising concerns within the Heart Team and judged as "arguable" for TF approach following angiography or CT-scan evaluation (hostile femoral access), with a RefD>/=5 mm and a MLD>/=3 mm.
7. Hostility score >/= 23 in at least one segment of the axis under evaluation.

Exclusion Criteria:

1. Life expectancy < 1 year
2. Subject has active infection requiring antibiotic therapy.
3. STS score ≥8%
4. Leriche syndrome or other forms of total occlusion of the aorta or both iliac axes.
5. Planned target limb major amputation (above the ankle).
6. History of prior endovascular or surgical procedure on the index limb within the past 30 days or planned within 30 days of the index procedure.
7. Subject in whom antiplatelet or anticoagulant therapy is contraindicated.
8. Subject has known allergy to contrast agents or medications used to perform endovascular intervention that cannot be adequately pre-treated.
9. Subject has known allergy to urethane, nylon, or silicone.
10. Subject is participating in another research study involving an investigational agent (pharmaceutical, biologic, or medical device) that has not reached the primary endpoint.
11. Subject has other medical, social or psychological problems that, in the opinion of the investigator, preclude them from receiving this treatment, and the procedures and evaluations pre- and post-treatment.
12. The use of specialty balloons, re-entry or atherectomy devices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with calcified ilio-femoral arteries eligible for trans-femoral TAVI
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-07-22 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility and safety on the trans-femoral (TF) approach | Index procedure - 1 Month
  Comparison of feasibility and safety on the TF approach as the composite of:
  * Valve implant unsuccess due to difficulties in advancing through the ilio-femoral vascular axe
  * Absence of cross over from PTA to IVL or vice-versa
  * Absence of severe vascular and bleeding complications at discharge and at 1 month follow up visit, as defined by VARC-3

SECONDARY OUTCOMES:
MAEs | Within 30 days after index procedure
  30-day composite occurrence of major clinical events: all-cause death, myocardial infarction and stroke
Vascular and bleeding complications | Within 30 days after index procedure
  30-day occurrence of vascular and bleeding complications according to the VARC-3 definition
Device-related vascular complication | Discharge, 1-months, 6-months
  Any device-related vascular complication
Residual stenosis, Degree of dissection, Final Flow | Index procedure
  Angiographic analysis from DSA
Procedural time duration, amount of contrast media and radiation dose. | Index procedure
  Procedural analysis
Centralized analysis of the angiographic parameters | Index procedure
  Centralized analysis of the angiographic parameters
Stent Implantation | Index procedure
  Need for stent implantation on the procedural vascular access axe.
Functional capacity of the inferior limbs | 6-months
  Functional capacity of the inferior limbs at 6 months.
Patency at the distal level of the vascular access site | 6-months
  Ultrasound defined patency at the distal level of the vascular access site after 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Ribichini, MD, PhD, Study Director — AOUI, Verona
Locations (5):
- Italy (5):
  - AOU Cardiology Ancona, Ancona
  - AULLS3 Cardiology Mestre, Mestre
  - AULSS2 Cardiology Treviso, Treviso
  - AOUI Cardiology Verona, Verona
  - AULLS8 Cardiology Vicenza, Vicenza

IPD SHARING:
Plan to Share IPD: No